CLINICAL TRIAL: NCT04488770
Title: A Double-Blind Randomized, Placebo-Controlled, Single and Repeated Oral Dose Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics (Including Food Effect) of GSK3882347 in Healthy Participants
Brief Title: Safety, Tolerability and Pharmacokinetic Investigation of GSK3882347 in Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 212148; 2020-000680-23 (EudraCT Number)
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-05

CONDITIONS: Urinary Tract Infections
Keywords: SAD; MAD; FTIH; Pharmacokinetics; Urinary Tract Infections; GSK3882347
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Part 1 will consist of two cohorts (Cohorts 1 and 2) with a maximum of four periods in a cross-over design conducted in two separate cohorts. Part 2 consists of a maximum of four ascending repeat-dose cohorts (Cohorts 3 to 6) for which participants, will receive a single oral dose of GSK3882347 or placebo for 7 days.
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study with participants and the site staff blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Part 1 (SAD) Cohort 1:Participants receiving GSK3882347 (Experimental): In this single ascending dose phase, participants will receive GSK3882347 50 milligram (mg), 150 mg and 250 mg orally on Day 1 of period 1, 2 and 3 respectively. Period 4 will be conducted to assess food effect based on the observed human PK.
  Interventions: Drug: GSK3882347
- Part 1 (SAD),Cohort 1:Participants receiving Placebo (Placebo Comparator): In this single ascending dose phase, participants will receive matching Placebo orally on Day 1 of period 1, 2 and 3. Period 4 will be conducted to assess food effect based on the observed human PK.
  Interventions: Drug: Placebo
- Part 1 (SAD),Cohort 2: Participants receiving GSK3882347 (Experimental): In this single ascending dose phase, participants will receive GSK3882347 500 mg, 15 mg and 900 mg orally on Day 1 of period 1, 3 and 2 respectively.
  Interventions: Drug: GSK3882347
- Part 1 (SAD),Cohort 2: Participants receiving Placebo (Placebo Comparator): In this single ascending dose phase, participants will receive matching Placebo orally on Day 1 of period 1, 3 and 2.
  Interventions: Drug: Placebo
- Part 2 (MAD),Cohort 3: Participants receiving GSK3882347 50mg (Experimental): In this multiple ascending dose phase, participants will receive GSK3882347 50 mg orally on Day 1 to Day 7 of the study. The dose to be administered may be changed based on clinical safety, tolerability and PK findings in Part 1.
  Interventions: Drug: GSK3882347
- Part 2 (MAD),Cohort 3: Participants receiving Placebo (Placebo Comparator): In this multiple ascending dose phase, participants will receive matching Placebo orally on Day 1 to Day 7 of the study.
  Interventions: Drug: Placebo
- Part 2 (MAD),Cohort 4: Participants receiving GSK3882347 150mg (Experimental): GSK3882347 150 mg will be administered orally to the participants on Day 1 to day 7 of the study. This is a projected dose. The dose administered in Part 2, Cohort 4 will be based on PK/PD results from preceding dosing cohorts.
  Interventions: Drug: GSK3882347
- Part 2 (MAD),Cohort 4: Participants receiving Placebo (Placebo Comparator): In this multiple ascending dose phase, participants will receive matching Placebo orally on Day 1 to Day 7 of the study.
  Interventions: Drug: Placebo
- Part 2(MAD),Cohort 5: Participants receiving GSK3882347 500mg (Experimental): GSK3882347 500 mg will be administered orally to the participants on Day 1 to day 7 of the study. This is a projected dose. The dose administered in Part 2, Cohort 5 will be based on PK/PD results from preceding dosing cohorts.
  Interventions: Drug: GSK3882347
- Part 2 (MAD),Cohort 5: Participants receiving Placebo (Placebo Comparator): In this multiple ascending dose phase, participants will receive matching Placebo orally on Day 1 to Day 7 of the study.
  Interventions: Drug: Placebo
- Part 2(MAD),Cohort 6: Participants receiving GSK3882347 900mg (Experimental): GSK3882347 900 mg will be administered orally to the participants on Day 1 to day 7 of the study. This is a projected dose. The dose administered in Part 2, Cohort 6 will be based on PK/PD results from preceding dosing cohorts.
  Interventions: Drug: GSK3882347
- Part 2(MAD),Cohort 6: Participants receiving Placebo (Placebo Comparator): In this multiple ascending dose phase, participants will receive matching Placebo orally on Day 1 to Day 7 of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3882347 — Capsule of 10-200mg dose strength will be provided in labelled High Density Polyethylene (HDPE) bottles.
  Arms: Part 1 (SAD) Cohort 1:Participants receiving GSK3882347; Part 1 (SAD),Cohort 2: Participants receiving GSK3882347; Part 2 (MAD),Cohort 3: Participants receiving GSK3882347 50mg; Part 2 (MAD),Cohort 4: Participants receiving GSK3882347 150mg; Part 2(MAD),Cohort 5: Participants receiving GSK3882347 500mg; Part 2(MAD),Cohort 6: Participants receiving GSK3882347 900mg
Drug: Placebo — Matching strength placebo capsules will be provided
  Arms: Part 1 (SAD),Cohort 1:Participants receiving Placebo; Part 1 (SAD),Cohort 2: Participants receiving Placebo; Part 2 (MAD),Cohort 3: Participants receiving Placebo; Part 2 (MAD),Cohort 4: Participants receiving Placebo; Part 2 (MAD),Cohort 5: Participants receiving Placebo; Part 2(MAD),Cohort 6: Participants receiving Placebo

SUMMARY:
This is a phase 1, 2-part, double-blind (sponsor-unblinded), randomized, placebo-controlled, first time in human (FTIH) study, that includes both single-ascending and multiple-ascending dose phase to assess the safety, tolerability, and pharmacokinetics (PK) of GSK3882347 in healthy adult men and Woman of Non Childbearing Potential (WONCBP). Part 1 will be the single ascending dose (SAD) phase and Part 2 will be the multiple ascending dose (MAD) phase. Each participant in the SAD cohort will receive a single dose of GSK3882347 or placebo (PBO) in 3:1 ratio and in Part 2 (MAD), participants will be randomized in a 4:1 ratio to receive active treatment and placebo. Part 1 will consist of two cohorts with a maximum of four-period for each cohort, the food effect evaluation will be conducted in last period (Period 4) in only one of the cohorts based on the observed human pharmacokinetics (PK). Part 2 will consist of maximum of four cohorts for each of the MAD dose or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring. A participant with a clinical abnormality or laboratory parameter(s) not specifically listed in the exclusion or exclusion criteria that is outside the reference range for the population being studied may be included only if the investigator, in consultation with the Medical Monitor (if required), agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Participants with Body weight at least 50.0 kilograms (kg) (110 pound [lbs]) for males and 45.0 kg (99 lbs.) for females; and body mass index (BMI) within the range 18.5 - 32.0 kilograms per meter square (kg/m^2) (inclusive).
* Male and female participants; a female participant is eligible to participate if she is of WONCBP; Male participants are eligible to participate if they agree to the following during the intervention period for at least five days, corresponding to time needed to eliminate study intervention(s) (e.g. 5 terminal half-lives) after the last dose of study intervention), refrain from donating sperm, be abstinent from heterosexual or homosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; must agree to use contraception/barrier, agree to use a male condom.
* Capable of giving signed informed consent as described in which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Participants with history or presence of cardiovascular, respiratory, hepatic, urological, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data
* Alanine transaminase (ALT) greater than 1.5 times upper limit of normal (ULN).
* Bilirubin greater than 1.5 times ULN (isolated bilirubin greater than1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin is less than 35%)
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (except for Gilbert's syndrome or asymptomatic gallstones).
* Medical history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome.
* Male participants with heart rate of less than 45 or greater than 100 beats per minute (bpm), females with less than 50 or greater than 100 bpm.
* Participants with PR interval less than 120 or greater than 220 milliseconds (msec); QRS duration less than 70 msec or greater than 120 msec; QTcF interval greater than 450 msec.
* Evidence of previous myocardial infarction on ECG (does not include ST segment changes associated with re-polarization).
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], Wolff-Parkinson-White [WPW] syndrome).
* Sinus Pauses greater than 3 seconds.
* Any significant arrhythmia which, in the opinion of the Investigator or GSK Medical Monitor, will interfere with the safety for the individual participant.
* Non-sustained or sustained ventricular tachycardia (3 consecutive ventricular ectopic beats).
* Current or history of renal disease, or estimated creatinine clearance <90 milliliter (mL)/minute/1.73meter^2 or serum creatinine greater than ULN at screening.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the first dose of study intervention, unless in the opinion of the Investigator and the GSK medical monitor, the medication will not interfere with the study procedures or compromise participant safety.
* Use of a systemic antimicrobial within 30 days of screening.
* Participation in the study would result in loss of blood or blood products in excess of 500 mL within 56 days.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation within the last 30 days before signing of consent in any other clinical study involving an investigational study intervention or any other type of medical research.
* Positive human immunodeficiency virus (HIV) antibody test.
* Presence of Hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention.
* Positive Hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Positive Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention.
* Positive pre-study drug/alcohol screen.
* Any history of substance abuse or a positive test for drugs of abuse at screening or admission.
* A positive highly sensitive pregnancy test (urine or serum as required by local regulations) at screening.
* A positive laboratory confirmation of COVID-19 infection, or high clinical index of suspicion for COVID-19.
* Part 1 (Food Effect): Participant must have no dietary restrictions (e.g., lactose intolerance) or inability to eat a high fat meal.
* Regular alcohol consumption within 6 months prior to the study defined as: An average weekly intake of greater than 21 units for males or greater than 14 units for females. One unit is equivalent to approximately (250 mL) of beer, (100 mL) of wine or (35 mL) measure of spirits.
* Positive smoke breathalyzer indicative of smoking history at screening and each in-house admission to the clinical research unit or regular use of tobacco- or nicotine-containing products (e.g. nicotine patches or vaporizing devices) within 6 months prior to screening.
* Hypersensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-part, first-time-in-human (FTIH), dose-escalation, placebo (PBO)-controlled, single dose (SD) (Part 1) and repeat dose (RD) (Part 2) study to determine the safety, tolerability and pharmacokinetic (PK) profile of GSK3882347 in healthy participants. The study was conducted at a single center in the United Kingdom.
Pre-assignment Details: A total of 61 participants (21 participants in Part 1 and 40 participants in Part 2) were enrolled in the study.
Groups:
- Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD 250 mg/SD PBO: Healthy participants in Part 1 Cohort 1 received a single dose (SD) of GSK3882347 50 milligrams (mg) on Day 1 in treatment Period 1, followed by a SD of GSK3882347 150 mg on Day 1 in treatment Period 2, followed by a SD of GSK3882347 250 mg on Day 1 in treatment Period 3, further followed by a SD of Placebo (PBO) on Day 1 in treatment Period 4. Cohort 1 was a 4-period cross-over.
- Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD PBO/SD 250mg Fed: Healthy participants in Part 1 Cohort 1 received a SD of GSK3882347 50 mg on Day 1 in treatment Period 1, followed by a SD of GSK3882347 150 mg on Day 1 in treatment Period 2, followed by a SD of PBO on Day 1 in treatment Period 3, further followed by a SD of GSK3882347 250 mg under fed condition on Day 1 in treatment Period 4. Cohort 1 was a 4-period cross-over.
- Part1-Cohort1: GSK3882347 SD 50mg/SD PBO/SD 250mg/SD 250mg Fed: Healthy participants in Part 1 Cohort 1 received a SD of GSK3882347 50 mg on Day 1 in treatment Period 1, followed by a SD of PBO on Day 1 in treatment Period 2, followed by a SD of GSK3882347 250 mg on Day 1 in treatment Period 3, further followed by a SD of GSK3882347 250 mg under fed condition on Day 1 in treatment Period 4. Cohort 1 was a 4-period cross-over.
- Part1-Cohort1:SD PBO/GSK3882347 SD 150mg/SD 250mg/SD 250mg Fed: Healthy participants in Part 1 Cohort 1 received a SD of PBO on Day 1 in treatment Period 1, followed by a SD of GSK3882347 150 mg on Day 1 in treatment Period 2, followed by a SD of GSK3882347 250 mg on Day 1 in treatment Period 3, further followed by a SD of GSK3882347 250 mg under fed condition on Day 1 in treatment Period 4. Cohort 1 was a 4-period cross-over.
- Part 1-Cohort 2: SD PBO/GSK3882347 SD 900 mg/SD 15 mg: Healthy participants in Part 1 Cohort 2 received a SD of PBO on Day 1 in treatment Period 1, followed by a SD of GSK3882347 900 mg on Day 1 in treatment Period 2, further followed by a SD of GSK3882347 15 mg on Day 1 in treatment Period 3. Cohort 2 was a 3-period cross-over.
- Part 1-Cohort 2: GSK3882347 SD 500 mg/SD PBO/SD 15 mg: Healthy participants in Part 1 Cohort 2 received a SD of GSK3882347 500 mg on Day 1 in treatment Period 1, followed by a SD of PBO on Day 1 in treatment Period 2, further followed by a SD of GSK3882347 15 mg on Day 1 in treatment Period 3. Cohort 2 was a 3-period cross-over.
- Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD PBO: Healthy participants in Part 1 Cohort 2 received a SD of GSK3882347 500 mg on Day 1 in treatment Period 1, followed by a SD of GSK3882347 900 mg on Day 1 in treatment Period 2, further followed by a SD of PBO on Day 1 in treatment Period 3. Cohort 2 was a 3-period cross-over.
- Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD 15 mg: Healthy participants in Part 1 Cohort 2 received a SD of GSK3882347 500 mg on Day 1 in treatment Period 1, followed by a SD of GSK3882347 900 mg on Day 1 in treatment Period 2, further followed by a SD of GSK3882347 15 mg on Day 1 in treatment Period 3. Cohort 2 was a 3-period cross-over.
- Part 2: Repeat Dose Placebo: Healthy participants in Part 2 received repeat dose (RD) of Placebo on Days 1 to 7.
- Part 2: Repeat Dose GSK3882347 50 mg: Healthy participants in Part 2 received RD of GSK3882347 50 mg on Days 1 to 7.
- Part 2: Repeat Dose GSK3882347 150 mg: Healthy participants in Part 2 received RD of GSK3882347 150 mg on Days 1 to 7.
- Part 2: Repeat Dose GSK3882347 500 mg: Healthy participants in Part 2 received RD of GSK3882347 500 mg on Days 1 to 7.
- Part 2: Repeat Dose GSK3882347 900 mg: Healthy participants in Part 2 received RD of GSK3882347 900 mg on Days 1 to 7.
Period: Part 1-Cohort 1: Period 1 (Up to 5 Days)
Arm/Group | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD 250 mg/SD PBO | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD PBO/SD 250mg Fed | Part1-Cohort1: GSK3882347 SD 50mg/SD PBO/SD 250mg/SD 250mg Fed | Part1-Cohort1:SD PBO/GSK3882347 SD 150mg/SD 250mg/SD 250mg Fed | Part 1-Cohort 2: SD PBO/GSK3882347 SD 900 mg/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD PBO/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD PBO | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD 15 mg | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1-Cohort 1: Period 2 (Up to 5 Days)
Arm/Group | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD 250 mg/SD PBO | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD PBO/SD 250mg Fed | Part1-Cohort1: GSK3882347 SD 50mg/SD PBO/SD 250mg/SD 250mg Fed | Part1-Cohort1:SD PBO/GSK3882347 SD 150mg/SD 250mg/SD 250mg Fed | Part 1-Cohort 2: SD PBO/GSK3882347 SD 900 mg/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD PBO/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD PBO | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD 15 mg | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Started | 2 | 2 | 2 | 2 (New participant enrolled and dosed as a replacement of withdrawn participant) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1-Cohort 1: Period 3 (Up to 5 Days)
Arm/Group | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD 250 mg/SD PBO | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD PBO/SD 250mg Fed | Part1-Cohort1: GSK3882347 SD 50mg/SD PBO/SD 250mg/SD 250mg Fed | Part1-Cohort1:SD PBO/GSK3882347 SD 150mg/SD 250mg/SD 250mg Fed | Part 1-Cohort 2: SD PBO/GSK3882347 SD 900 mg/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD PBO/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD PBO | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD 15 mg | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1-Cohort 1: Period 4 (Up to 5 Days)
Arm/Group | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD 250 mg/SD PBO | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD PBO/SD 250mg Fed | Part1-Cohort1: GSK3882347 SD 50mg/SD PBO/SD 250mg/SD 250mg Fed | Part1-Cohort1:SD PBO/GSK3882347 SD 150mg/SD 250mg/SD 250mg Fed | Part 1-Cohort 2: SD PBO/GSK3882347 SD 900 mg/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD PBO/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD PBO | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD 15 mg | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Started | 2 (New participant enrolled and dosed as a replacement of withdrawn participant) | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1-Cohort 2: Period 1 (Up to 5 Days)
Arm/Group | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD 250 mg/SD PBO | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD PBO/SD 250mg Fed | Part1-Cohort1: GSK3882347 SD 50mg/SD PBO/SD 250mg/SD 250mg Fed | Part1-Cohort1:SD PBO/GSK3882347 SD 150mg/SD 250mg/SD 250mg Fed | Part 1-Cohort 2: SD PBO/GSK3882347 SD 900 mg/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD PBO/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD PBO | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD 15 mg | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Started | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1-Cohort 2: Period 2 (Up to 5 Days)
Arm/Group | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD 250 mg/SD PBO | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD PBO/SD 250mg Fed | Part1-Cohort1: GSK3882347 SD 50mg/SD PBO/SD 250mg/SD 250mg Fed | Part1-Cohort1:SD PBO/GSK3882347 SD 150mg/SD 250mg/SD 250mg Fed | Part 1-Cohort 2: SD PBO/GSK3882347 SD 900 mg/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD PBO/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD PBO | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD 15 mg | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Started | 0 | 0 | 0 | 0 | 2 | 2 (New participant enrolled and dosed as a replacement of withdrawn participant) | 2 (New participant enrolled and dosed as a replacement of withdrawn participant) | 2 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1-Cohort 2: Period 3 (Up to 5 Days)
Arm/Group | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD 250 mg/SD PBO | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD PBO/SD 250mg Fed | Part1-Cohort1: GSK3882347 SD 50mg/SD PBO/SD 250mg/SD 250mg Fed | Part1-Cohort1:SD PBO/GSK3882347 SD 150mg/SD 250mg/SD 250mg Fed | Part 1-Cohort 2: SD PBO/GSK3882347 SD 900 mg/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD PBO/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD PBO | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD 15 mg | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Started | 0 | 0 | 0 | 0 | 2 (New participant enrolled and dosed as a replacement of withdrawn participant) | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Up to 26 Days)
Arm/Group | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD 250 mg/SD PBO | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD PBO/SD 250mg Fed | Part1-Cohort1: GSK3882347 SD 50mg/SD PBO/SD 250mg/SD 250mg Fed | Part1-Cohort1:SD PBO/GSK3882347 SD 150mg/SD 250mg/SD 250mg Fed | Part 1-Cohort 2: SD PBO/GSK3882347 SD 900 mg/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD PBO/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD PBO | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD 15 mg | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD 250 mg/SD PBO | Part1-Cohort1:GSK3882347 SD 50mg/SD 150mg/SD PBO/SD 250mg Fed | Part1-Cohort1: GSK3882347 SD 50mg/SD PBO/SD 250mg/SD 250mg Fed | Part1-Cohort1:SD PBO/GSK3882347 SD 150mg/SD 250mg/SD 250mg Fed | Part 1-Cohort 2: SD PBO/GSK3882347 SD 900 mg/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD PBO/SD 15 mg | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD PBO | Part 1-Cohort 2: GSK3882347 SD 500 mg/SD 900 mg/SD 15 mg | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg | Total
Number analyzed (Participants) | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 2 | 8 | 8 | 8 | 8 | 8 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 2 | 8 | 8 | 8 | 8 | 8 | 61
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 2 | 8 | 8 | 8 | 8 | 8 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 5
  Asian- South East Asian Heritage | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
  White- White/Caucasian/European Heritage | 3 | 2 | 1 | 2 | 3 | 2 | 3 | 2 | 6 | 8 | 6 | 7 | 6 | 51
  Mixed race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Number of participants with common (greater than or equal to [>=]5 percent [%]) non-serious AEs is presented.
Time Frame: Up to 3 months
Population: Safety Population comprised of all participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Single Dose Placebo: Healthy participants in Part 1 received a SD of Placebo on Day 1 in either treatment Periods 1, 2, 3 and 4.
- Part 1: Single Dose GSK3882347 15 mg: Healthy participants in Part 1 received a SD of GSK3882347 15 mg on Day 1 in treatment Period 3.
- Part 1: Single Dose GSK3882347 50 mg: Healthy participants in Part 1 received a SD of GSK3882347 50 mg on Day 1 in treatment Period 1.
- Part 1: Single Dose GSK3882347 150 mg: Healthy participants in Part 1 received a SD of GSK3882347 150 mg on Day 1 in treatment Period 2.
- Part 1: Single Dose GSK3882347 250 mg: Healthy participants in Part 1 received a SD of GSK3882347 250 mg on Day 1 in treatment Period 3.
- Part 1: Single Dose GSK3882347 250 mg Fed: Healthy participants in Part 1 received a SD of GSK3882347 250 mg under fed condition on Day 1 in treatment Period 4.
- Part 1: Single Dose GSK3882347 500 mg: Healthy participants in Part 1 received a SD of GSK3882347 500 mg on Day 1 in treatment Period 1.
- Part 1: Single Dose GSK3882347 900 mg: Healthy participants in Part 1 received a SD of GSK3882347 900 mg on Day 1 in treatment Period 2.
Arm/Group | Part 1: Single Dose Placebo | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Non-serious AEs | 7 | 1 | 2 | 2 | 3 | 2 | 3 | 2
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 2: Number of Participants With Non-serious AEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Number of participants with common (>=5%) non-serious AEs is presented.
Time Frame: Up to 26 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Participants
  Non-serious AEs | 5 | 4 | 2 | 7 | 7
  SAEs | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Part 1: Number of Participants With Treatment Related AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Number of participants with treatment related AEs is presented.
Time Frame: Up to 3 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Single Dose Placebo | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part 2: Number of Participants With Treatment Related AEs
Description: as for outcome 3
Time Frame: Up to 26 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Participants | 1 | 2 | 0 | 0 | 0

5. Primary Outcome: Part 1: Number of Participants With Worst-case Hematology Results Relative to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected to analyze hematocrit,hemoglobin,leukocytes,lymphocytes,neutrophils and platelets. PCI ranges were <0.075 or >0.54 proportion of red blood cells in blood for hematocrit, <25 or >180 grams per liter(g/L) for hemoglobin,<3 or >20 x10^9 cells per liter(cells/L) for leukocytes,<0.8 x10^9 cells/L for lymphocytes,<1.5 x10^9 cells/L for neutrophils and <100 or >550 x10^9 cells/L for platelets.Participants were counted in worst case category that their value changes to(low,within range or no change or high),unless there is no change in their category.Participants whose laboratory value category was unchanged(for example[e.g.],High to High),or whose value became within range, were recorded in"To within Range or No Change" category.Participants were counted twice if the participant has values that changed 'To Low' and 'To High',so the percentages may not add to 100%.Baseline=latest pre-dose assessment with a non-missing value, including those from unscheduled visits
Time Frame: Up to 3 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Single Dose Placebo | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Hematocrit: To Low | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 1
  Hematocrit: To within Range or No Change | 12 | 4 | 6 | 6 | 5 | 5 | 5 | 5
  Hematocrit: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Hemoglobin: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Leukocytes: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Lymphocytes: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Neutrophils: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Platelets: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part 2: Number of Participants With Worst-case Hematology Results Relative to PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected to analyze hematocrit,hemoglobin,leukocytes,lymphocytes,neutrophils and platelets. PCI ranges were <0.075 or >0.54 proportion of red blood cells in blood for hematocrit, <25 or >180 grams per liter(g/L) for hemoglobin,<3 or >20 x10^9 cells per liter(cells/L) for leukocytes,<0.8 x10^9 cells/L for lymphocytes,<1.5 x10^9 cells/L for neutrophils and <100 or >550 x10^9 cells/L for platelets.Participants were counted in worst case category that their value changes to(low,within range or no change or high),unless there is no change in their category.Participants whose laboratory value category was unchanged(e.g.,High to High),or whose value became within range, were recorded in"To within Range or No Change" category.Participants were counted twice if the participant has values that changed 'To Low' and 'To High',so the percentages may not add to 100%.Baseline=latest pre-dose assessment with a non-missing value, including those from unscheduled visits
Time Frame: Up to 26 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Participants
  Hematocrit: To Low | 2 | 2 | 1 | 0 | 1
  Hematocrit: To within Range or No Change | 6 | 6 | 7 | 8 | 7
  Hematocrit: To High | 0 | 0 | 0 | 0 | 0
  Hemoglobin: To Low | 0 | 1 | 0 | 0 | 0
  Hemoglobin: To within Range or No Change | 8 | 7 | 8 | 8 | 8
  Hemoglobin: To High | 0 | 0 | 0 | 0 | 0
  Leukocytes: To Low | 1 | 0 | 0 | 0 | 0
  Leukocytes: To within Range or No Change | 7 | 8 | 8 | 8 | 8
  Leukocytes: To High | 0 | 0 | 0 | 0 | 0
  Lymphocytes: To Low | 0 | 0 | 0 | 0 | 0
  Lymphocytes: To within Range or No Change | 8 | 8 | 8 | 8 | 8
  Lymphocytes: To High | 0 | 0 | 0 | 0 | 0
  Neutrophils: To Low | 0 | 0 | 1 | 0 | 0
  Neutrophils: To within Range or No Change | 8 | 8 | 7 | 8 | 8
  Neutrophils: To High | 0 | 0 | 0 | 0 | 0
  Platelets: To Low | 0 | 0 | 0 | 0 | 0
  Platelets: To within Range or No Change | 8 | 8 | 8 | 8 | 8
  Platelets: To High | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Part 1: Number of Participants With Worst-case Clinical Chemistry Results Relative to PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected to analyze PCI ranges: >=2 times Upper limit of Normal(ULN) Units per Liter(U/L) for Alanine aminotransferase(ALT),>=2 times ULN U/L for alkaline phosphatase(ALP), >=2 times ULN U/L for aspartate aminotransferase(AST),>=1.5 times ULN micromoles/L for bilirubin,<2 or >2.75 millimoles/L (mmol/L) for calcium,<3 or >9 mmol/L for glucose,<3 or >5.5 mmol/L for potassium and <130 or >150 mmol/L for sodium.Participants were counted in worst case category that their value changes to(low,within range or no change or high),unless there is no change in their category.Participants whose laboratory value category was unchanged(e.g.,High to High),or whose value became within range,were recorded in"To within Range or No Change" category.Participants were counted twice if the participant has values that changed 'To Low' and 'To High',so the percentages may not add to 100%.Baseline=latest pre-dose assessment with a non-missing value,including those from unscheduled visits
Time Frame: Up to 3 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Single Dose Placebo | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  ALT: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  ALT: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALP: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALP: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  ALP: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  AST: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Bilirubin: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Calcium: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Glucose: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Potassium: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Sodium: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Part 2: Number of Participants With Worst-case Clinical Chemistry Results Relative to PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected to analyze PCI ranges: >=2 times ULN U/L for Alanine aminotransferase(ALT),>=2 times ULN U/L for alkaline phosphatase(ALP), >=2 times ULN U/L for aspartate aminotransferase(AST),>=1.5 times ULN micromoles/L for bilirubin,<2 or >2.75 mmol/L for calcium,<3 or >9 mmol/L for glucose,<3 or >5.5 mmol/L for potassium and <130 or >150 mmol/L for sodium.Participants were counted in worst case category that their value changes to(low,within range or no change or high),unless there is no change in their category.Participants whose laboratory value category was unchanged(e.g.,High to High),or whose value became within range,were recorded in"To within Range or No Change" category.Participants were counted twice if the participant has values that changed 'To Low' and 'To High',so the percentages may not add to 100%.Baseline=latest pre-dose assessment with a non-missing value,including those from unscheduled visits.
Time Frame: Up to 26 days
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Participants
  ALT: To Low | 0 | 0 | 0 | 0 | 0
  ALT: To within Range or No Change | 8 | 8 | 8 | 8 | 8
  ALT: To High | 0 | 0 | 0 | 0 | 0
  ALP: To Low | 0 | 0 | 0 | 0 | 0
  ALP: To within Range or No Change | 8 | 8 | 8 | 8 | 8
  ALP: To High | 0 | 0 | 0 | 0 | 0
  AST: To Low | 0 | 0 | 0 | 0 | 0
  AST: To within Range or No Change | 8 | 8 | 8 | 8 | 8
  AST: To High | 0 | 0 | 0 | 0 | 0
  Bilirubin: To Low | 0 | 0 | 0 | 0 | 0
  Bilirubin:To within Range or No Change | 7 | 8 | 8 | 8 | 8
  Bilirubin: To High | 1 | 0 | 0 | 0 | 0
  Calcium: To Low | 0 | 0 | 0 | 0 | 0
  Calcium: To within Range or No Change | 8 | 8 | 8 | 8 | 8
  Calcium: To High | 0 | 0 | 0 | 0 | 0
  Glucose: To Low: number analyzed (Participants) | 4 | 8 | 8 | 0 | 0
  Glucose: To Low | 0 | 0 | 0 |  |
  Glucose: To within Range or No Change: number analyzed (Participants) | 4 | 8 | 8 | 0 | 0
  Glucose: To within Range or No Change | 4 | 8 | 8 |  |
  Glucose: To High: number analyzed (Participants) | 4 | 8 | 8 | 0 | 0
  Glucose: To High | 0 | 0 | 0 |  |
  Potassium: To Low | 0 | 0 | 0 | 0 | 0
  Potassium:To within Range or No Change | 8 | 8 | 8 | 8 | 8
  Potassium: To High | 0 | 0 | 0 | 0 | 0
  Sodium: To Low | 0 | 0 | 0 | 0 | 0
  Sodium: To within Range or No Change | 8 | 8 | 8 | 8 | 8
  Sodium: To High | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Part 1: Number of Participants With Worst Case Urinalysis Results Post Baseline Relative to Baseline
Description: Urine samples were collected for the analysis of urine parameters including occult blood and protein by dipstick. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as no change/decreased, increase to positive for urine occult blood and protein indicating proportional concentrations in the urine sample. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Number of participants with worst case urinalysis results Post Baseline relative to Baseline is presented.
Time Frame: Up to 3 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Single Dose Placebo | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Occult Blood, No change/decreased | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 5
  Occult blood, Increase to positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Protein, No change/decreased | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Protein, Increase to positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Part 2: Number of Participants With Worst Case Urinalysis Results Post Baseline Relative to Baseline
Description: Urine samples were collected for the analysis of urine parameters including occult blood and protein by dipstick. The dipstick test gave results in a semi-quantitative manner (proportional concentrations in urine samples), and results for urinalysis parameters were recorded as no change/decreased, increase to positive for urine occult blood and protein. 'No change/decreased' indicates no change from Baseline results or decreased in results from Baseline including change in negative results. 'Increase to positive' indicates increase in result from Baseline. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Number of participants with worst case urinalysis results Post Baseline relative to Baseline is presented.
Time Frame: Up to 26 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Participants
  Occult Blood, No change/decreased | 8 | 8 | 7 | 8 | 8
  Occult blood, Increase to positive | 0 | 0 | 1 | 0 | 0
  Protein, No change/decreased | 7 | 8 | 8 | 8 | 8
  Protein, Increase to trace | 1 | 0 | 0 | 0 | 0

11. Primary Outcome: Part 1: Number of Participants With Worst Case Vital Signs Results Relative to PCI Criteria Post Baseline Relative to Baseline
Description: Vital signs were assessed including Systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate (PR). PCI ranges were <85 (Low), 85-160 (Normal) and >160 (High) for SBP; <45 (Low), 45-100 (Normal), >100 (High) for DBP; <40 (Low), 40-110 (Normal), >110 (High) for pulse rate. Participants were counted in worst case category that their value changes to(low,within range or no change, high),unless there is no change in their category.Participants whose laboratory value category was unchanged(e.g.,High to High),or whose value became within range, were recorded in"To within Range or No Change" category.Participants were counted twice if the participant has values that changed 'To Low' and 'To High',so the percentages may not add to 100%.Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits
Time Frame: Up to 3 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Single Dose Placebo | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  SBP: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  SBP: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  DBP: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR: To within Range or No Change | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  PR: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Part 2: Number of Participants With Worst Case Vital Signs Results Relative to PCI Criteria Post Baseline Relative to Baseline
Description: as for outcome 11
Time Frame: Up to 26 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Participants
  SBP: To Low | 0 | 0 | 0 | 0 | 0
  SBP: To within Range or No Change | 8 | 8 | 8 | 8 | 8
  SBP: To High | 0 | 0 | 0 | 0 | 0
  DBP: To Low | 0 | 0 | 0 | 0 | 0
  DBP: To within Range or No Change | 8 | 8 | 8 | 8 | 8
  DBP: To High | 0 | 0 | 0 | 0 | 0
  PR: To Low | 1 | 0 | 1 | 0 | 0
  PR: To within Range or No Change | 7 | 8 | 7 | 8 | 8
  PR: To High | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Part 1: Number of Participants With Worst Case Abnormal Electrocardiogram (ECG) Results Post Baseline Relative to Baseline
Description: A 12-lead ECG was recorded with the participant in a semi-supine position after a rest of at least 10 minutes. Twelve lead ECGs were obtained by using an automated ECG machine that measured PR, QRS, QT, and corrected QT (QTc) intervals and calculated heart rate. Data for abnormal not clinically significant (NCS) and clinically significant (CS) ECG findings are presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Up to 3 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Single Dose Placebo | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Abnormal: NCS | 3 | 1 | 1 | 0 | 0 | 2 | 1 | 1
  Abnormal: CS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Part 2: Number of Participants With Worst Case Abnormal ECG Results Post Baseline Relative to Baseline
Description: as for outcome 13
Time Frame: Up to 26 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Participants
  Abnormal: NCS | 3 | 3 | 6 | 6 | 3
  Abnormal: CS | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero to 24 Hours (AUC[0-24]) After Single Dose Administration of GSK3882347
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK3882347. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16 and 24 hours post-dose in each treatment period
Population: PK Population comprised of all participants in the safety population who had at least 1 non-missing PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours*nanograms per milliliter | 1671.7 (20.9) | 6514.1 (12.3) | 17717.9 (18.0) | 28472.2 (27.9) | 21456.4 (7.8) | 48381.2 (26.9) | 65150.2 (28.3)

16. Primary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC[0-t]) After Single Dose Administration of GSK3882347
Description: Blood samples were collected at indicated time points for PK analysis of GSK3882347. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours*nanograms per milliliter | 1954.3 (24.7) | 8249.8 (18.2) | 22266.9 (16.9) | 36561.0 (26.7) | 29091.9 (10.6) | 63052.2 (26.1) | 88901.9 (31.8)

17. Primary Outcome: Part 1: Area Under the Concentration-time Curve Extrapolated From Time Zero to Infinity (AUC[0-infinity]) After Single Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours*nanograms per milliliter | 2167.0 (23.4) | 8425.5 (18.1) | 22433.7 (16.8) | 36768.0 (26.5) | 29316.1 (10.5) | 63377.3 (26.1) | 89424.5 (32.1)

18. Primary Outcome: Part 1: Maximum Plasma Concentration (Cmax) After Single Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Nanograms per milliliter | 165.7 (22.3) | 661.7 (14.8) | 1825.8 (21.2) | 3126.7 (31.3) | 1834.5 (13.4) | 4671.3 (27.4) | 5771.6 (24.6)

19. Primary Outcome: Part 1: Plasma Concentrations at 24 Hours (C24h) After Single Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16 and 24 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Nanograms per milliliter | 27.32 (29.7) | 106.70 (39.5) | 283.18 (24.7) | 500.35 (28.8) | 453.82 (13.6) | 853.98 (35.0) | 1291.37 (41.0)

20. Primary Outcome: Part 1: Time to Cmax (Tmax) After Single Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose in each treatment period
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 3.000 [2.00 to 4.00] | 4.000 [2.00 to 4.18] | 4.000 [2.00 to 6.00] | 4.000 [2.00 to 6.00] | 4.000 [2.00 to 8.00] | 4.000 [2.00 to 4.00] | 4.000 [2.00 to 8.00]

21. Primary Outcome: Part 1: Lag Time for Absorption (Tlag) After Single Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose in each treatment period
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 0.375 [0.25 to 0.50] | 0.250 [0 to 0.50] | 0.250 [0 to 0.50] | 0.250 [0 to 0.25] | 0.250 [0.25 to 1.50] | 0.250 [0.25 to 0.50] | 0.250 [0.25 to 0.50]

22. Primary Outcome: Part 1: Terminal Elimination Half-life (T1/2) After Single Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 11.407 (17.7) | 12.269 (14.5) | 11.538 (10.1) | 12.277 (16.0) | 12.984 (10.3) | 12.630 (11.6) | 12.690 (13.8)

23. Primary Outcome: Part 2: Area Under the Concentration-time Curve Over the Dosing Interval Tau (AUC[0-tau]) After Repeat Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Days 1 and 7: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
Hours*nanograms per milliliter
  Day 1 | 5862.9 (16.2) | 20191.4 (25.6) | 45400.0 (38.8) | 53753.9 (27.8)
  Day 7 | 6144.9 (8.7) | 21109.5 (27.9) | 61202.0 (27.4) | 82351.1 (22.7)

24. Primary Outcome: Part 2: Cmax After Repeat Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Days 1 and 7: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
Nanograms per milliliter
  Day 1 | 586.0 (20.8) | 2179.1 (29.5) | 4409.4 (34.2) | 4933.1 (24.0)
  Day 7 | 600.4 (21.9) | 2007.4 (31.7) | 5370.3 (21.2) | 6575.2 (28.6)

25. Primary Outcome: Part 2: Tmax After Repeat Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Days 1 and 7: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
Hours
  Day 1 | 4.000 [2.00 to 6.00] | 3.000 [1.50 to 4.00] | 4.000 [4.00 to 6.00] | 4.008 [4.00 to 6.00]
  Day 7 | 4.000 [2.00 to 6.00] | 4.000 [2.00 to 6.00] | 4.000 [2.00 to 6.00] | 4.000 [2.00 to 6.00]

26. Primary Outcome: Part 2: Plasma Concentrations Over the Dosing Interval (Ctau) After Repeat Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Days 1 and 7: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
Nanograms per milliliter
  Day 1 | 90.98 (46.8) | 292.53 (22.2) | 789.85 (46.7) | 1084.55 (31.8)
  Day 7 | 109.28 (26.8) | 368.34 (29.7) | 1170.62 (39.2) | 1864.47 (23.1)

27. Primary Outcome: Part 1: Urine Concentration Between 22-24 Hours (C22-24) After Single Dose Administration of GSK3882347
Description: Urine samples were collected at indicated time points for PK analysis of GSK3882347. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Day 1: 22-24 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Micrograms per milliliter | 1.55 (71.3) | 2.99 (95.9) | 11.27 (146.7) | 15.26 (133.9) | 11.42 (148.0) | 48.54 (161.8) | 33.50 (75.0)

28. Primary Outcome: Part 2: Urine Concentration Between 22-24 Hours (C22-24) After Repeat Dose Administration of GSK3882347
Description: as for outcome 27
Time Frame: Day 1 and Day 7: 22-24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
Micrograms per milliliter
  Day 1 | 2.95 (52.5) | 11.98 (64.8) | 18.15 (42.8) | 38.43 (90.6)
  Day 7 | 2.56 (84.4) | 16.50 (26.7) | 23.60 (69.6) | 57.15 (75.2)

29. Primary Outcome: Part 1: Amount of Drug Excreted in Urine of Unchanged Drug (Ae Total) After Single Dose Administration of GSK3882347
Description: as for outcome 27
Time Frame: At 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-22, 22-24, 24-26, 26-32, 32-38, 38-48, 48-60, 60-72, 72-84, 84-96 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Milligrams | 11.16 (15.7) | 32.01 (9.4) | 106.86 (25.5) | 146.43 (20.5) | 95.17 (9.2) | 306.93 (20.8) | 430.03 (22.5)

30. Primary Outcome: Part 2: Amount of Drug Excreted in Urine of Unchanged Drug (Ae Total) After Repeat Dose Administration of GSK3882347
Description: as for outcome 27
Time Frame: Days 1 and 7: At 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-22, 22-24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
Milligrams
  Day 1 | 24.77 (17.6) | 88.30 (14.2) | 188.49 (32.5) | 267.16 (18.4)
  Day 7 | 26.71 (19.0) | 108.20 (17.4) | 258.08 (18.7) | 390.10 (13.0)

31. Primary Outcome: Part 1: Percentage of the Given Dose of Drug Excreted in Urine (%fe Total) After Single Dose Administration of GSK3882347
Description: Urine samples were collected at indicated time points for PK analysis of GSK3882347. PK parameters were analyzed using standard non-compartmental analysis. %fe was calculated as: (Ae total/Dose)*100 percent (%).
Time Frame: as for outcome 29
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent dose excreted
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Percent dose excreted | 74.43 (15.7) | 64.02 (9.4) | 71.24 (25.5) | 58.57 (20.5) | 38.07 (9.2) | 61.39 (20.8) | 47.78 (22.5)

32. Primary Outcome: Part 2: Percentage of the Given Dose of Drug Excreted in Urine (%fe Total) After Single Dose Administration of GSK3882347
Description: Urine samples were collected at indicated time points for PK analysis of GSK3882347. PK parameters were analyzed using standard non-compartmental analysis. %fe was calculated as: (Ae total/Dose)*100%.
Time Frame: Day 1 and Day 7: At 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-22, 22-24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent dose excreted
Arm/Group | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
Percent dose excreted
  Day 1 | 49.54 (17.6) | 58.87 (14.2) | 37.70 (32.5) | 29.68 (18.4)
  Day 7 | 53.42 (19.0) | 72.13 (17.4) | 51.62 (18.7) | 43.34 (13.0)

33. Primary Outcome: Part 1: Renal Clearance of Drug (CLr) After Single Dose Administration of GSK3882347
Description: Urine samples were collected at indicated time points for PK analysis of GSK3882347. PK parameters were analyzed using standard non-compartmental analysis. CLr was calculated as: Ae total/AUC(0-t)
Time Frame: as for outcome 29
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Liters per hour | 5.71 (31.7) | 3.88 (25.8) | 4.80 (30.9) | 4.00 (19.1) | 3.27 (14.2) | 4.87 (17.5) | 4.84 (22.7)

34. Primary Outcome: Part 2: Renal Clearance of Drug (CLr) After Repeat Dose Administration of GSK3882347
Description: as for outcome 33
Time Frame: Day 1 and Day 7: At 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-22, 22-24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
Liters per hour
  Day 1 | 4.24 (20.8) | 4.38 (28.6) | 4.16 (28.7) | 4.98 (19.1)
  Day 7 | 4.34 (16.9) | 5.12 (19.8) | 4.22 (28.6) | 4.73 (18.0)

35. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero to 12 Hours (AUC[0-12]) After Single Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8 and 12 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours*nanogram per milliliter | 1181.6 (20.3) | 4609.1 (10.2) | 12519.7 (19.7) | 20127.1 (29.1) | 14009.0 (10.1) | 33030.8 (26.8) | 42353.5 (26.6)

36. Secondary Outcome: Part 1: Plasma Concentrations at 12 Hours (C12) After Single Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8 and 12 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Nanograms per milliliter | 58.73 (26.7) | 232.96 (17.1) | 636.41 (18.5) | 947.62 (27.5) | 857.73 (9.5) | 1806.50 (33.9) | 2714.12 (43.9)

37. Secondary Outcome: Part 1: Apparent Oral Clearance (CL/F) After Single Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Liters per hour | 6.92 (23.4) | 5.93 (18.1) | 6.69 (16.8) | 6.80 (26.5) | 8.53 (10.5) | 7.89 (26.1) | 10.06 (32.1)

38. Secondary Outcome: Part 1: Apparent Volume of Distribution After Oral Administration (Vz/F) After Single Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Liters | 113.92 (22.8) | 105.04 (6.7) | 111.30 (22.7) | 120.43 (34.3) | 159.74 (11.3) | 143.76 (30.1) | 184.26 (24.1)

39. Secondary Outcome: Part 1: Mean Residence Time (MRT) After Single Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose in each treatment period
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 15.775 [12.76 to 23.46] | 16.843 [12.45 to 19.61] | 15.614 [13.38 to 19.62] | 16.262 [14.36 to 19.84] | 18.818 [16.57 to 20.73] | 17.259 [15.41 to 19.89] | 18.630 [15.32 to 22.90]

40. Secondary Outcome: Part 2: Area Under the Concentration-time Curve From Time Zero to 12 Hours (AUC[0-12]) After Repeat Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Days 1 and 7: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8 and 12 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
Hours*nanogram per milliliter
  Day 1 | 4076.3 (16.4) | 14411.9 (28.9) | 30660.3 (37.1) | 35231.6 (26.3)
  Day 7 | 4222.8 (11.0) | 14506.3 (28.9) | 41187.1 (24.1) | 53121.9 (23.9)

41. Secondary Outcome: Part 2: Plasma Concentrations at 12 Hours (C12) After Repeat Dose Administration of GSK3882347
Description: as for outcome 16
Time Frame: Days 1 and 7: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8 and 12 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
Nanograms per milliliter
  Day 1 | 214.4 (23.5) | 709.1 (19.9) | 1704.8 (42.1) | 2068.2 (36.0)
  Day 7 | 221.5 (11.8) | 776.1 (28.3) | 2360.8 (30.6) | 3218.5 (21.6)

42. Secondary Outcome: Part 1: Dose Proportionality of GSK3882347 for Dose Levels 15 mg to 900 mg Using AUC(0-infinity) After Single Dose Administration of GSK3882347 Under Fasted Condition
Description: Blood samples were collected at indicated time points for PK analysis of GSK3882347. PK parameters were analyzed using standard non-compartmental analysis. Dose proportionality was assessed using Power model. Log-e(dose) was fitted as fixed effect and participant was fitted as random effect. Kenward and Roger method and unstructured covariance structure was used. Slope and 90% confidence interval (CI) for the slope are presented. The SD 250 mg fed treatment was not considered in the analysis.
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose in each treatment period
Population: PK Population. Only those participants with data available at the specified data points were analyzed. The dose proportionality was assessed for doses administered under fasted conditions only. Being a FTIH study, the impact of food on drug PK was unknown; hence it would have been inaccurate to include fed arm in dose proportionality assessment in this FTIH study. Therefore, 250 mg fed arm was not considered in dose proportionality assessment
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Groups:
- Part 1: GSK3882347 SD 15 mg to 900 mg: Healthy participants were administered single dose of GSK3882347 15 mg, 50 mg, 150 mg, 250 mg, 500 mg and 900 mg under fasted condition in either of treatment Period 1, 2, 3 or 4 according to randomization schedule
Arm/Group | Part 1: GSK3882347 SD 15 mg to 900 mg
Number analyzed (Participants) | 19
Slope of log dose | 0.919 [0.889 to 0.949]

43. Secondary Outcome: Part 1: Dose Proportionality of GSK3882347 for Dose Levels 15 mg to 900 mg Using Cmax After Single Dose Administration of GSK3882347 Under Fasted Condition
Description: Blood samples were collected at indicated time points for PK analysis of GSK3882347. PK parameters were analyzed using standard non-compartmental analysis. Dose proportionality was assessed using Power model. Log-e(dose) was fitted as fixed effect and participant was fitted as random effect. Kenward and Roger method and unstructured covariance structure was used. Slope and 90% CI for the slope are presented. The SD 250 mg fed treatment was not considered in the analysis.
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose in each treatment period
Population: as for outcome 42
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | Part 1: GSK3882347 SD 15 mg to 900 mg
Number analyzed (Participants) | 19
Slope of log dose | 0.903 [0.865 to 0.941]

44. Secondary Outcome: Part 2: Dose Proportionality of GSK3882347 for Dose Levels 50 mg to 900 mg Using AUC(0-tau) After Repeat Dose Administration of GSK3882347
Description: Blood samples were collected at indicated time points for PK analysis of GSK3882347. PK parameters were analyzed using standard non-compartmental analysis. Dose proportionality was assessed using Power model. Log-e(dose) was fitted as fixed effect and participant was fitted as random effect. Kenward and Roger method and unstructured covariance structure was used. Slope and 90% CI for the slope are presented.
Time Frame: Day 1 and Day 7: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Groups:
- Part 2: GSK3882347 RD 50 mg to 900 mg: Participants were administered repeat dose of GSK3882347 50 mg, 150 mg, 500 mg or 900 mg
Arm/Group | Part 2: GSK3882347 RD 50 mg to 900 mg
Number analyzed (Participants) | 32
Slope of log dose
  Day 1 | 0.770 [0.684 to 0.857]
  Day 7 | 0.908 [0.841 to 0.976]

45. Secondary Outcome: Part 2: Dose Proportionality of GSK3882347 for Dose Levels 50 mg to 900 mg Using Cmax After Repeat Dose Administration of GSK3882347
Description: as for outcome 44
Time Frame: Day 1 and Day 7: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | Part 2: GSK3882347 RD 50 mg to 900 mg
Number analyzed (Participants) | 32
Slope of log dose
  Day 1 | 0.736 [0.644 to 0.829]
  Day 7 | 0.841 [0.763 to 0.920]

46. Secondary Outcome: Part 2: Observed Accumulation Ratio (Ro) Using AUC(0-tau) After Repeat Dose Administration of GSK3882347
Description: Blood samples were collected at indicated time points for PK analysis of GSK3882347. PK parameters were analyzed using standard non-compartmental analysis. Accumulation ratio was calculated as AUC(0-tau) at Day 7 divided by AUC(0-tau) at Day 1 for GSK3882347. Mixed effect model was used to assess accumulation ratio for the log transformed parameters. Treatment, day and the interaction of treatment and day were fitted as fixed effect. Participant was fitted as random effect. Kenward and Roger method and unstructured covariance structure was used.
Time Frame: Day 1 and Day 7: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24 hours post-dose
Population: PK Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
Ratio | 1.05 [0.93 to 1.18] | 1.05 [0.93 to 1.18] | 1.35 [1.20 to 1.52] | 1.53 [1.36 to 1.72]

47. Secondary Outcome: Part 2: Time Invariance of GSK3882347
Description: Blood samples were collected at indicated time points for the analysis of time invariance. Time invariance was calculated as AUC(0-tau) at Day 7 divided by AUC(0-infinity) at Day 1 for GSK3882347. Mixed effect ANOVA model was used to assess time invariance for the log transformed parameters. Treatment, day and the interaction of treatment and day were fitted as fixed effect. Participant was fitted as random effect. Kenward and Roger method and unstructured covariance structure was used.
Time Frame: Day 1 and Day 7: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24 hours post-dose
Population: PK Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
Ratio | 0.83 [0.74 to 0.94] | 0.87 [0.77 to 0.99] | 1.07 [0.95 to 1.20] | 1.13 [1.00 to 1.28]

48. Secondary Outcome: Part 2: Pre-dose Plasma Concentrations After Repeat Dose Administration of GSK3882347 From Days 3 to 7
Description: Blood samples were collected at indicated time points for PK analysis of GSK3882347.
Time Frame: Days 3, 4, 5, 6 and 7: Pre-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
Nanograms per milliliter
  Day 3: Pre-dose | 99.48 (19.360) | 326.89 (81.306) | 1157.589 (432.3864) | 1578.14 (328.085)
  Day 4: Pre-dose | 96.66 (16.722) | 344.56 (112.891) | 1212.368 (438.9076) | 1883.90 (560.646)
  Day 5: Pre-dose | 96.16 (15.683) | 329.37 (88.100) | 1166.770 (369.9656) | 1724.07 (524.054)
  Day 6: Pre-dose | 97.50 (21.275) | 339.83 (100.604) | 1157.068 (384.6052) | 1776.54 (513.638)
  Day 7: Pre-dose | 92.46 (14.390) | 300.16 (75.925) | 1105.470 (464.5923) | 1769.40 (618.929)

49. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero to 24 Hours (AUC[0-24]) After Single Dose Administration of GSK3882347 250 mg Under Fasted and Fed Conditions for Assessment of Food Effect
Description: Blood samples were collected at indicated time points for PK analysis of GSK3882347 250 mg under fasted and fed conditions for assessment of food effect. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Standard Error); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed
Number analyzed (Participants) | 6 | 6
Hours*nanogram per milliliter | 28472.2 (0.08) | 21456.4 (0.08)
Statistical Analysis 1: Comparison: Part 1: Single Dose GSK3882347 250 mg vs Part 1: Single Dose GSK3882347 250 mg Fed; Test type: Other; Ratio of Geometric Mean = 0.75, 90% CI 2-sided [0.61 to 0.93] — Mixed Effect Model has been used to assess Food Effect for the log transformed parameter AUC(0-24). Treatment in the fed/fasted state is fitted as Fixed Effect. Participant is fitted as Random Effect. Unstructured covariance structure is used

50. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC [0-t]) After Single Dose Administration of GSK3882347 250 mg Under Fasted and Fed Conditions for Assessment of Food Effect
Description: as for outcome 49
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Standard Error); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed
Number analyzed (Participants) | 6 | 6
Hours*nanogram per milliliter | 36561.0 (0.08) | 29091.9 (0.08)
Statistical Analysis 1: Comparison: Part 1: Single Dose GSK3882347 250 mg vs Part 1: Single Dose GSK3882347 250 mg Fed; Test type: Other; Ratio of Geometric Mean = 0.80, 90% CI 2-sided [0.65 to 0.98] — Mixed Effect Model was used to assess Food Effect for the log transformed parameter AUC(0-t). Treatment in the fed/fasted state was fitted as Fixed Effect. Participant was fitted as Random Effect. Unstructured covariance structure was used

51. Secondary Outcome: Part 1: Area Under the Concentration-time Curve Extrapolated From Time Zero to Infinity (AUC [0-infinity]) After Single Dose Administration of GSK3882347 250 mg Under Fasted and Fed Conditions for Assessment of Food Effect
Description: as for outcome 49
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Standard Error); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed
Number analyzed (Participants) | 6 | 6
Hours*nanogram per milliliter | 36768.0 (0.08) | 29316.1 (0.08)
Statistical Analysis 1: Comparison: Part 1: Single Dose GSK3882347 250 mg vs Part 1: Single Dose GSK3882347 250 mg Fed; Test type: Other; Ratio of Geometric Mean = 0.80, 90% CI 2-sided [0.65 to 0.98] — Mixed Effect Model was used to assess Food Effect for log transformed parameter AUC(0-infinity). Treatment in the fed/fasted state was fitted as Fixed Effect. Participant was fitted as Random Effect. Unstructured covariance structure was used

52. Secondary Outcome: Part 1: Maximum Plasma Concentration (Cmax) After Single Dose Administration of GSK3882347 250 mg Under Fasted and Fed Conditions for Assessment of Food Effect
Description: as for outcome 49
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Standard Error); unit: Nanograms per milliliter
Arm/Group | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed
Number analyzed (Participants) | 6 | 6
Nanograms per milliliter | 3126.7 (0.10) | 1834.5 (0.10)
Statistical Analysis 1: Comparison: Part 1: Single Dose GSK3882347 250 mg vs Part 1: Single Dose GSK3882347 250 mg Fed; Test type: Other; Ratio of Geometric Mean = 0.59, 90% CI 2-sided [0.46 to 0.75] — Mixed Effect Model was used to assess Food Effect for the log transformed parameter Cmax. Treatment in the fed/fasted state was fitted as Fixed Effect. Participant was fitted as Random Effect. Unstructured covariance structure was used

53. Secondary Outcome: Part 1: Plasma Concentrations at 24 Hours (C24h) After Single Dose Administration of GSK3882347 250 mg Under Fasted and Fed Conditions for Assessment of Food Effect
Description: as for outcome 49
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Standard Error); unit: Nanograms per milliliter
Arm/Group | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed
Number analyzed (Participants) | 6 | 6
Nanograms per milliliter | 494.7 (0.09) | 449.2 (0.09)
Statistical Analysis 1: Comparison: Part 1: Single Dose GSK3882347 250 mg vs Part 1: Single Dose GSK3882347 250 mg Fed; Test type: Other; Ratio of Geometric Mean = 0.91, 90% CI 2-sided [0.74 to 1.11] — Mixed Effect Model was used to assess Food Effect for the log transformed parameter C24h. Treatment in the fed/fasted state was fitted as Fixed Effect. Participant was fitted as Random Effect. Unstructured covariance structure was used

54. Secondary Outcome: Part 1: Tmax After Single Dose Administration of GSK3882347 250 mg Under Fasted and Fed Conditions for Assessment of Food Effect
Description: as for outcome 49
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed
Number analyzed (Participants) | 6 | 6
Hours | 4.000 [2.00 to 6.00] | 4.000 [2.00 to 8.00]
Statistical Analysis 1: Comparison: Part 1: Single Dose GSK3882347 250 mg vs Part 1: Single Dose GSK3882347 250 mg Fed; Test type: Other; Median Difference (Net) = 0.000, 90% CI 2-sided [0.000 to 2.000] — Wilcoxon matched pair test was used to assess Food Effect for the parameter Tmax

55. Secondary Outcome: Part 1: Tlag After Single Dose Administration of GSK3882347 250 mg Under Fasted and Fed Conditions for Assessment of Food Effect
Description: as for outcome 49
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 32, 48, 72 and 96 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed
Number analyzed (Participants) | 6 | 6
Hours | 0.250 [0 to 0.25] | 0.250 [0.25 to 1.50]
Statistical Analysis 1: Comparison: Part 1: Single Dose GSK3882347 250 mg vs Part 1: Single Dose GSK3882347 250 mg Fed; Test type: Other; Median Difference (Net) = 0.000, 90% CI 2-sided [0.000 to 0.250] — Wilcoxon matched pair test was used to assess Food Effect for the parameter Tlag

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs and Non-SAEs were collected from the start of study treatment up to 3 months for Part 1 and up to 26 days for Part 2
Description: All-cause mortality, SAEs and Non-SAEs were reported for the Safety Population which comprised of all participants who received at least one dose of study treatment.
Arm/Group | Part 1: Single Dose Placebo | Part 1: Single Dose GSK3882347 15 mg | Part 1: Single Dose GSK3882347 50 mg | Part 1: Single Dose GSK3882347 150 mg | Part 1: Single Dose GSK3882347 250 mg | Part 1: Single Dose GSK3882347 250 mg Fed | Part 1: Single Dose GSK3882347 500 mg | Part 1: Single Dose GSK3882347 900 mg | Part 2: Repeat Dose Placebo | Part 2: Repeat Dose GSK3882347 50 mg | Part 2: Repeat Dose GSK3882347 150 mg | Part 2: Repeat Dose GSK3882347 500 mg | Part 2: Repeat Dose GSK3882347 900 mg
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/14 | 1/6 | 2/6 | 2/6 | 3/6 | 2/6 | 3/6 | 2/6 | 5/8 | 4/8 | 2/8 | 7/8 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Single Dose Placebo (N=14) | Part 1: Single Dose GSK3882347 15 mg (N=6) | Part 1: Single Dose GSK3882347 50 mg (N=6) | Part 1: Single Dose GSK3882347 150 mg (N=6) | Part 1: Single Dose GSK3882347 250 mg (N=6) | Part 1: Single Dose GSK3882347 250 mg Fed (N=6) | Part 1: Single Dose GSK3882347 500 mg (N=6) | Part 1: Single Dose GSK3882347 900 mg (N=6) | Part 2: Repeat Dose Placebo (N=8) | Part 2: Repeat Dose GSK3882347 50 mg (N=8) | Part 2: Repeat Dose GSK3882347 150 mg (N=8) | Part 2: Repeat Dose GSK3882347 500 mg (N=8) | Part 2: Repeat Dose GSK3882347 900 mg (N=8)
Headache (Nervous system disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site vesicles (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Product use complaint (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT04488770/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT04488770/SAP_001.pdf